CLINICAL TRIAL: NCT06257160
Title: Superiority Randomized Controlled Trial of Ultrasound-guided PENG Block Compared to Surgical Infiltration in the Analgesia of Posterior Total Hip Arthroplasty Surgery
Acronym: PENGORINF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PO24003
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hip Arthropathy; Hip Arthrosis
Keywords: Analgesia; Hip; Arthroplasty; PENG; locoregional anesthesia; infiltration
MeSH Terms: conditions — Osteoarthritis, Hip; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical infiltration (Active Comparator)
  Interventions: Procedure: Surgical infiltration
- PENG Block ultrasound-guided (Experimental)
  Interventions: Procedure: PENG Block ultrasound-guided

INTERVENTIONS:
Procedure: Surgical infiltration — During surgery, local anesthetics are injected as follow: in the deep plane and in the subcutaneous territory.
  Infiltration of the deep plane corresponds to pericotyloid injection, with particular attention to the posterior subcapsular area, the obturator foramen and the psoas muscle. Infiltration of the muscular planes is added, with infiltration of the gluteal and pelvitrochanteric muscles.
  Arms: Surgical infiltration
Procedure: PENG Block ultrasound-guided — We perform the femoral block under ultrasound after anesthesia (general or rachianesthesia). The PENG block is a peripheral diffusion nerve block that specifically targets the articular divisions of the femoral, obturator and accessory obturator nerves.
  The femoral nerve innervates the four parts of the joint capsule, with inconsistency in the anterior inferomedial part of the capsule.
  The obturator nerve innervates the inferior part of the anterior face of the capsule.
  The accessory obturator nerve innervates the medial half of the hip joint capsule in over 50% of cases.
  Arms: PENG Block ultrasound-guided

SUMMARY:
Pain after total hip replacement (THR) surgery is severe. The target population is elderly and comorbid. Level III analgesics are responsible for significant side effects in this population. Locoregional analgesia, by reducing the consumption of painkillers, is an effective way of reducing morphine or morphine agonist consumption in this surgery. Furthermore, these techniques fit in perfectly with the objectives of accelerated rehabilitation after surgery. Surgical infiltration is a frequently used and effective analgesic technique. PENG block is a new locoregional anesthesia technique which initial results show promising analgesic efficacy and the absence of loss of strength through motor block.

In February 2022, we carried out a survey of national anesthetic practices in posterior hip arthroplasty, with the help of the SFAR (Société Française d'Anesthésie-Réanimation).

It shows that, despite the lack of plentiful literature on the subject, the PENG block is currently the most frequently performed pre-operative block in hip arthroplasty (PENG block in 39.5% of cases, femoral block in 13% of cases).

The survey also shows that in 41.5% of cases, no block is performed, and only intraoperative surgical infiltration is carried out.

PENG block and surgical infiltration are therefore the two analgesic techniques most frequently used in France today.

It is for these reasons that we feel it is essential to carry out a study comparing these two techniques.

DETAILED DESCRIPTION:
The aim of this study was to compare the clinical efficacy of these two locoregional analgesia strategies in posterior total hip replacement surgery: ultrasound-guided PENG block and surgical infiltration.

The study is a superiority randomized, double-blind (patient and evaluator will be blinded to the randomization group), single-center trial.

Two groups of patients will be compared: a group of patients benefiting from the echo-guided PENG block strategy, and a group of patients benefiting from intraoperative surgical infiltration.

The type of treatment (PENG block or surgical infiltration) will be randomized. The target population concerns patients scheduled for posterior total hip replacement surgery at Reims University Hospital If the hypothesis of the superior efficacy of echo-guided block PENG is confirmed, our analgesia strategy for total hip replacement surgery will be modified, enabling us to offer the most effective locoregional analgesia technique and thus reduce the morbidity and mortality associated with morphine consumption.

This could have both a medical and an economic impact, by optimizing post-operative monitoring and convalescence for these patients.

ELIGIBILITY:
Inclusion criteria:

* Patients eligible for posterior total hip replacement surgery at Reims University Hospital
* Patients agreeing to take part in the research and having signed the informed consent form
* Patients of full age
* Patients affiliated to a social security scheme

Exclusion criteria:

* Minor patients
* Patients protected by law
* Pregnant and breast-feeding women
* Patients with allergy to local anesthetics
* Patients with neuropathy
* Patients with an ASA score greater than or equal to 4
* Patients undergoing revision surgery on a total hip prosthesis
* Patients undergoing anterior total hip replacement surgery
* Patients suffering from a femur fracture
* Patients with a contraindication to Peng block.
* Patients refusing one of the proposed techniques.
* Persons deprived of their liberty by judicial or administrative decision.
* Persons under psychiatric care
* Persons unable to express their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | At 24 hours postoperative

SECONDARY OUTCOMES:
Pain evaluation | At 1 hour postoperative
  Numeric pain intensity scale
Pain evaluation | At 2 hours postoperative
  Numeric pain intensity scale
Pain evaluation | At 6 hours postoperative
  Numeric pain intensity scale
Pain evaluation | At 12 hours postoperative
  Numeric pain intensity scale
Pain evaluation | At 24 hours postoperative
  Numeric pain intensity scale
Pain evaluation | At 36 hours postoperative
  Numeric pain intensity scale
Pain evaluation | At 48 hours postoperative
  Numeric pain intensity scale
Success or failure at first stand up test | At 4 hours postoperative
Need for analgesia rescue technique | At 24 hours postoperative
10 meters walk test | At 24 hours postoperative
Muscle strength test | At 24 hours postoperative
Length of hospital stay | At the end of the stay
Adverse events due to consumption of morphine | At 24 hours postoperative
Adverse events due to PENG block ou surgical infiltration | At 24 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France